CLINICAL TRIAL: NCT03968523
Title: Loco/Regional Anaesthesia Evaluation in Laparoscopic Hernioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3467
Record Dates: First submitted 2019-05-20; First posted 2019-05-30 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Laparoscopic inguinal hernioplasty; TAP block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two randomized cohorts of treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each patient will be included in one cohort of treatment by a randomized criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Active Comparator): TAP block technique.
  Interventions: Procedure: TAP block
- Novel local infiltration technique (Experimental): Local analgesic infiltration in the mesh fixation site
  Interventions: Procedure: Novel local infiltration technique

INTERVENTIONS:
Procedure: Novel local infiltration technique — Local analgesic infiltration in the mesh fixation site
  Arms: Novel local infiltration technique
Procedure: TAP block — TAP block technique
  Arms: TAP block

SUMMARY:
Laparoscopic hernioplasty is associated with lesser postoperative pain and quick return to work. TAP block is the gold standard technique in this type of hernioplasty. Our aim is to compare TAP block with a novel local infiltration technique that uses direct laparoscopical vision.

DETAILED DESCRIPTION:
Laparoscopic hernioplasty is associated with lesser postoperative pain and quick return to work. TAP block is the gold standard technique in this type of hernioplasty. Our aim is to compare TAP block with a novel local infiltration technique that uses direct laparoscopical vision. Patients will be randomized into two arms of intervention that will be compared by a blind analysis. Primary outcomes will be postoperative pain evaluated systematically until 30 days postoperative, and analgesic consumption.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more.
* Programmed inguinal laparoscopic hernioplasty

Exclusion Criteria:

* Allergic to medication prescribed
* Story of mesh rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 30 days postoperative
  Postoperative main measured by an visual analogue scale

SECONDARY OUTCOMES:
Analgesics consumption | 30 days postoperative
  Time to analgesic consumption
type of analgesic consumption | 30 days
  type of analgesic consumption
pain at the moment of need of analgesics take | 30 days
  pain measured at the analgesic consumption

OTHER OUTCOMES:
Postoperative complications | 30 days postoperative
  Seroma, hematoma, surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Bertone, MD, Principal Investigator — Surgeon
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liem MS, van der Graaf Y, van Steensel CJ, Boelhouwer RU, Clevers GJ, Meijer WS, Stassen LP, Vente JP, Weidema WF, Schrijvers AJ, van Vroonhoven TJ. Comparison of conventional anterior surgery and laparoscopic surgery for inguinal-hernia repair. N Engl J Med. 1997 May 29;336(22):1541-7. doi: 10.1056/NEJM199705293362201. PMID 9164809
- [Background] Grant AM, Scott NW, O'Dwyer PJ; MRC Laparoscopic Groin Hernia Trial Group. Five-year follow-up of a randomized trial to assess pain and numbness after laparoscopic or open repair of groin hernia. Br J Surg. 2004 Dec;91(12):1570-4. doi: 10.1002/bjs.4799. PMID 15515112
- [Background] Joshi GP, Rawal N, Kehlet H; PROSPECT collaboration; Bonnet F, Camu F, Fischer HB, Neugebauer EA, Schug SA, Simanski CJ. Evidence-based management of postoperative pain in adults undergoing open inguinal hernia surgery. Br J Surg. 2012 Feb;99(2):168-85. doi: 10.1002/bjs.7660. Epub 2011 Sep 16. PMID 21928388
- [Background] Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. No abstract available. PMID 18020088
- [Background] Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. PMID 21154380
- See also: Comparison of conventional anterior surgery and laparoscopic surgery for inguinal-hernia repair. N Engl J M — https://www.ncbi.nlm.nih.gov/pubmed/9164809
- See also: Grant AM, Scott NW, O'Dwyer PJ; MRC Laparoscopic Groin Hernia Trial Group. Five-year follow-up of a randomized trial to assess pain and numbness after laparoscopic or open repair of groin hernia. Br J Surg. 2004 Dec;91(12):1570-4. — https://www.ncbi.nlm.nih.gov/m/pubmed/15515112/
- See also: Evidence-based management of postoperative pain in adults undergoing open inguinal hernia surgery. Br J Surg. 2012 Feb;99(2):168-85. d — https://www.ncbi.nlm.nih.gov/pubmed/21928388
- See also: Hebbard P, Fujiwara Y, Shibata Y, Royse C. Ultrasound-guided transversus abdominis plane (TAP) block. Anaesth Intensive Care. 2007 Aug;35(4):616-7. — https://www.ncbi.nlm.nih.gov/pubmed/18020088
- See also: Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. Review. — https://www.ncbi.nlm.nih.gov/pubmed/21154380